CLINICAL TRIAL: NCT01050907
Title: Treatment of Mucocutaneous Leishmaniasis With Miltefosine
Brief Title: Miltefosine to Treat Mucocutaneous Leishmaniasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Knight Therapeutics (USA) Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBL-MILT-201
Record Dates: First submitted 2010-01-12; First posted 2010-01-18 (Estimated); Results first posted 2020-09-30 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-08

CONDITIONS: Mucosal Leishmaniasis; Cutaneous Leishmaniasis
Keywords: leishmaniasis; cutaneous disease; mucosal disease; miltefosine
MeSH Terms: conditions — Leishmaniasis, Mucocutaneous; Leishmaniasis, Cutaneous; Leishmaniasis | interventions — miltefosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Miltefosine (Experimental): 2.5 mg/kg/day for 28 days
  Interventions: Drug: Miltefosine

INTERVENTIONS:
Drug: Miltefosine — 2.5 mg/kg/day for 28 days
  Other Names: Impavido

SUMMARY:
The purpose of this Treatment Investigational New Drug application was to make miltefosine available for mucocutaneous leishmaniasis patients presenting in the United States.

If entrance criteria were met, subjects with mucosal or cutaneous leishmaniasis received miltefosine at a targeted dose of 2.5 mg/kg/day for 28 days. During treatment at weeks 1, 2, and 4, the patient returned to the treatment facility to be assessed for adverse events. Blood for transaminase and creatinine values were drawn at the midpoint and at the end of therapy.

Patients returned to the treatment facility to be examined clinically at 6 weeks (ie, 2 weeks after the end of therapy), 3 months (2 months after therapy), and 7 months (6 months after treatment) for mucosal leishmaniasis and cutaneous leishmaniasis patients, and also at 13 months (12 months after treatment) for mucosal leishmaniasis patients.

DETAILED DESCRIPTION:
Subjects with mucosal leishmaniasis or cutaneous leishmaniasis from which Leishmania have already been identified were potentially eligible to be treated with miltefosine via this protocol. Treating Physicians with potentially eligible subjects contacted the protocol Principal Investigator (PI), and received the case report forms (CRF) from the PI. The Treating Physician completed the screening CRF pages for demographics, medical history, leishmaniasis history, clinical laboratory results that were available, and identification of Leishmania in the lesion, and sent the completed CRF pages to the PI. If after PI review, the subject was potentially eligible for the protocol, the PI sent the protocol, the miltefosine package insert, the informed consent form, and a blank copy of FDA form 1572 to the Treating Physician. Although this protocol would have already been approved by a "central" Institutional Review Board (IRB), if there was an additional need to have the Treating Physician's local IRB approve the protocol, the Treating Physician would obtain the approval, and obtain informed consent from the subject. The rest of the laboratory tests were accomplished so that all screening laboratory tests were completed prior to enrolling a potential subject. If in the physician's opinion the subject appeared eligible for enrollment, the Treating Physician sent to the PI the local IRB signature page (if needed), protocol signature page, informed consent signed by both the subject and the Treating Physician, the rest of the completed CRF pages for screening, and the form 1572 completed with the Treating Physician's information plus the Treating Physician's curriculum vitae. After the PI's review of these forms, the investigational product was sent from the drug repository to the Treating Physician for that subject's use.

Treatment was daily for 28 consecutive days. During treatment at weeks 1, 2, and 4, the subject returned to the treatment facility to be assessed for adverse events and to receive additional supply of medication if needed. Compliance with drug administration was assessed by subject interview and pill count. Blood for transaminase and creatinine values were drawn at the midpoint and at the end of therapy.

Subjects returned to the treatment facility to be examined clinically at Study Week 6, Study Months 3 and 7 months for mucosal leishmaniasis and cutaneous leishmaniasis subjects, and also at Study Month 13 for mucosal leishmaniasis subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Is the subject a male or female at least 18 years of age?
2. Does the subject weigh at least 30 kg?
3. Does the subject have a diagnosis of mucosal leishmaniasis or cutaneous leishmaniasis in at least one lesion by at least one of the following methods: 1) positive culture for promastigotes of lesion material, 2) microscopic identification of amastigotes in stained lesion tissue, 3) Polymerase chain reaction of lesion material?
4. In the opinion of the investigator, is the subject capable of understanding and complying with the protocol?
5. If female and of child-bearing potential, did the subject have a negative pregnancy test during screening and agree to use an acceptable method of birth control during the treatment phase and for 6 months after treatment is completed?
6. Has the patient signed informed consent?

Exclusion Criteria:

1. Is the subject a female who is breast-feeding?
2. Does the subject have a clinically significant medical disorder?

   * Thrombocyte count <100 x 10e9/L
   * Leukocyte count <3 x 10e9/L
   * Haemoglobin <10 g/100 mL
   * Aspartate transaminiase (ASAT), alanine transaminase (ALAT) >2 times upper limit of normal range
   * Bilirubin >1.5 times upper limit of normal range
   * Serum creatinine >1.5 times upper limit of normal range
   * Major surgery within last 2 weeks
   * Any non-compensated or uncontrolled condition
3. In the last 4 weeks up to the present, has the subject received other treatment for leishmaniasis, including any medication with pentavalent antimony; amphotericin B, paromomycin, or imidazoles?

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-05; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Berman, MD, Principal Investigator — Fast Track Drugs and Biologics LLC
Locations (2):
- United States (2):
  - For this treatment IND, each Physician entered patients at his/her own facility. Below data is for protocol central contact:, Bethesda, Maryland
  - NIH, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Miltefosine
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Miltefosine
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Cure of Lesions
Description: Percent of participants with clinical cure of all lesions. Ulcerated CL lesions were measured for the longest diameter and perpendicular width of ulceration; non-ulcerated lesions were measured for length and width of the raised area. A healed lesion was 100% reduction in lesion area (0x0); a cured lesion was a lesion healed at the Month 7 visit. For subjects with ML, an Ear, Nose, and Throat specialist examined the nasal and oral mucosa. Each site (nasal skin, nasal mucosa, palate, pharynx, larynx) was evaluated for signs of disease (erythema, edema, infiltration, erosion) and graded on a scale: 0=no disease, 1=mild disease, 2=moderate disease, 3=severe disease. Max score was 60 = poor outcome. Clinical response measured as a composite score, the mucosal severity score, which was the sum of the severity scores for each clinical sign at each clinical site of disease. A healed lesion had a score of 0 in absolute value (0% of the entrance score), and clinical cure was lesion is healed.
Time Frame: Week 6, Month 3, Month 7, and Month 13
Population: The evaluable population included all subjects who received daily doses of investigational product for at least 25 of the total of 28 days, had lesion measurements at Month 7 for cutaneous leishmaniasis or the month 13 visit for mucosal leishmaniasis, and who did not receive rescue medications to treat leishmaniasis at any time during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Miltefosine
Number analyzed (Participants) | 4
Participants | 3

2. Primary Outcome: Number of Participants With Adverse Events
Description: The number of participants with adverse events (AEs) by occurrence and severity. The Treating Physician monitored participants for the occurrence of AEs from the time the first investigational product was taken on Day 1 through the end of follow up at Month 7 for CL or Month 13 for ML. For the period between Study Day 1 and Study Week 6 (2 weeks after the end of therapy), all AEs regardless of seriousness or relationship to the investigational product were to be recorded on the case report form (CRF). For the period Week 6 to Month 7 for CL, or Month 13 for ML, only AEs requiring medical attention were recorded on the CRF.
Time Frame: Up to 7 months for CL; Up to 13 months for ML
Population: The safety population included all subjects who received any administration of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Miltefosine
Number analyzed (Participants) | 4
Participants | 4

ADVERSE EVENTS:
Time Frame: Up to 7 months for CL; Up to 13 months for ML
Arm/Group | Miltefosine
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Miltefosine (N=4)
Epididymitis (Reproductive system and breast disorders) | 1 (1)
Abdominal Pain Lower (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (7)
Vomiting (Gastrointestinal disorders) | 2 (8)
Rash Pruritic (Skin and subcutaneous tissue disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2010-03-06): https://cdn.clinicaltrials.gov/large-docs/07/NCT01050907/Prot_SAP_000.pdf